CLINICAL TRIAL: NCT04203810
Title: Effectiveness and Tolerability of Ectoin® Mouth and Throat Spray Althaea Honey (ERS09) Compared to Saline Spray in Patients Suffering From Sore Throat Due to Acute Pharyngitis and Dry Cough
Brief Title: Effectiveness and Tolerability of Ectoin® Mouth and Throat Spray Althaea Honey (ERS09)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: btph-044-2019-ERS09
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2020-07

CONDITIONS: Sore Throat; Acute Pharyngitis; Cough
MeSH Terms: conditions — Pharyngitis; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ectoin® Mouth and Throat Spray Althaea Honey (Experimental): 4 puffs to be administered as needed several times a day for patients aged ≥ 12 years. A maximum of 10 applications per day should not be exceeded.
  Interventions: Device: Ectoin® Mouth and Throat Spray Althaea Honey (ERS09)
- EMSER® Hals- und Rachenspray (throat spray) (Active Comparator): 1 to 3 puffs to be administered several times a day
  Interventions: Device: EMSER® Hals-und Rachenspray (throat spray)

INTERVENTIONS:
Device: Ectoin® Mouth and Throat Spray Althaea Honey (ERS09) — 4 puffs to be administered as needed several times a day for patients aged ≥ 12 years. A maximum of 10 applications per day should not be exceeded.
  Arms: Ectoin® Mouth and Throat Spray Althaea Honey
Device: EMSER® Hals-und Rachenspray (throat spray) — 1 to 3 puffs to be administered several times a day
  Arms: EMSER® Hals- und Rachenspray (throat spray)

SUMMARY:
The aim of this multicentre, actively controlled, randomized, open label, parallel group, prospective, comparator study is to collect data on the clinical effectiveness and tolerability of the medical device ERS09 compared to a well-established comparator spray in the symptomatic treatment of sore throat due to acute pharyngitis and dry cough.

DETAILED DESCRIPTION:
The aim of this study is to collect data on the clinical effectiveness and tolerability of Ectoin® Mouth and Throat Spray Althaea Honey (ERS09) compared to the well-established comparator spray EMSER® Hals- und Rachenspray (both medical devices) in the symptomatic treatment of sore throat due to acute pharyngitis and dry cough.

The principle mode of action of ectoine is based on the physical interaction of the compatible solute with water and the resulting stabilizing effects of the ectoine hydro complex on the epithelial tissue treated. Althaea has so-called mucilaginous effects, that means generally a shielding of the irritated mucus membranes by thin polysaccharide layers. Such mucilaginous polymer layers lead to rehydration, coating of peripheral sensory receptors, and therefore to a reduction of throat irritation and dry coughing. Honey acts predominantly as demulcent with its viscous liquid constitution based on mainly fructose and glucose. The combination of all three substances may result in a multi-modal treatment of the symptoms of sore throat and dry cough.

Patients will be randomly assigned to one of the following treatment groups:

* treatment with ERS09
* treatment with comparator (EMSER® Hals- und Rachenspray)

Patients' symptoms will be documented by the physician in investigator questionnaires at visits 1, 2 and 3. At visit 1 the patients will receive a patient diary for daily documentation of their symptoms. In addition, patients and investigators will be asked to evaluate the overall effectiveness and tolerability of ERS09 spray at visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign and date an Informed Consent consistent with International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP)/ISO14155 guidelines and local regulation prior to participation in the trial
* Individuals regardless of gender 12 years old or older
* Patients with sore throat due to acute pharyngitis and dry cough, both with an onset of symptoms no more than 72 hours prior to Visit 1
* Sore Throat Pain Intensity Score ≥ 40 mm (measured on a 100 mm visual analogue scale [VAS])

Exclusion Criteria:

* Hypersensitivity to Ectoin, Althaea off., Honey or any of the other ingredients of the ERS09 or the comparator
* Fructose intolerance or glucose-galactose malabsorption
* Pregnant or breast-feeding women
* Suspected bacterial pharyngitis
* Individuals younger than 12 years
* Symptoms since more than 72 hours
* Use of any pain or cough medication (i.e. analgesic/ anti-pyretic/ anti-inflammatory or mucolytic/ expectorant/ antitussive) within 24 hours preceding enrolment in the study
* Oral lesions or oral surgical procedures within 1 month prior to enrolment in the study
* Patients for who the Investigator believes will not comply with the study protocol (e.g. patients with drug abuse or with a history of a serious psychiatric disorder as well as patients unwilling to give informed consent or to abide by the requirements of the protocol)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Change of mean total symptom score | 7 days
  Baseline adjusted mean change of patient's assessment of total symptom score (patient diary) averaged over 7 treatment days
Change of daily symptom score | 1 day
  Baseline adjusted daily change of patient's assessment of total symptom score (patient diary)

SECONDARY OUTCOMES:
Adverse events (AE) and serious adverse events (SAE) during treatment phase | 7 +/- 2 days
  Evaluation of severity, nature and frequency of AEs/SAEs and their relationship to the investigational devices

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Moesges, Prof. Dr., Principal Investigator — ClinCompetence GmbH, Genter Str. 7, 50672 Cologne, Germany
Locations (12):
- Germany (12):
  - Dr. Pasch, Aachen
  - Dr. Sondermann, Aachen
  - Dr. Männer, Arnsberg
  - Dr. Kienle-Gogolok, Bad Schönborn
  - Dr. Ginko, Bonn
  - Dr. Vent, Cologne
  - Praxis für Hals-Nasen-Ohren-Heilkunde, Dresden
  - Dr. Thieme, Duisburg
  - Dr. Horn, Heidelberg
  - Dr. Lenzenhuber, Jülich
  - Dr. Konzelmann, Röthenbach
  - Reiber, Schorndorf

IPD SHARING:
Plan to Share IPD: No